CLINICAL TRIAL: NCT04028492
Title: VP-VLY-686-3301: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase Iii Study To Assess The Efficacy Of Tradipitant In Relieving Symptoms Of Gastroparesis
Brief Title: Evaluating the Safety and Efficacy of Tradipitant vs. Placebo in Idiopathic and Diabetic Gastroparesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-3301
Record Dates: First submitted 2019-07-10; First posted 2019-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Gastroparesis; Diabetic Gastroparesis; Gastroparesis
Keywords: gastroparesis; idiopathic; diabetic; tradipitant; nausea; vomiting; stomach; motility; functional; NK-1 antagonist; neurokinin 1 receptor; substance p
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tradipitant (Experimental): Oral Capsule
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator): Oral Capsule
  Interventions: Drug: Placebo
- Open Label Tradipitant (Experimental): Oral Capsule
  Interventions: Drug: Open Label Tradipitant

INTERVENTIONS:
Drug: Tradipitant — BID
  Arms: Tradipitant
Drug: Placebo — BID
  Arms: Placebo
Drug: Open Label Tradipitant — BID
  Arms: Open Label Tradipitant

SUMMARY:
To investigate the safety and efficacy of tradipitant versus placebo in relieving nausea and other symptoms of gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastroparesis
* Demonstrated delayed gastric emptying
* Presence of moderate to severe nausea
* Body Mass Index (BMI) of ≥18 and ≤40 kg/m2

Exclusion Criteria:

* Another active disorder or treatment which could explain or contribute to symptoms of gastroparesis
* A positive test for drugs of abuse at the screening or evaluation visits;
* Exposure to any investigational medication in the past 60 days
* Gastrectomy, fundoplication, vagotomy, pyloroplasty, bariatric surgery, or gastric stimulation device surgically implanted within the last year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in daily average nausea severity scores from the Gastroparesis Core Symptom Daily Diary (GCS-DD) | 12 weeks
  A daily symptom diary asking patients to rate their nausea on a Likert scale from 0-5 (0=none, 5= very severe).

SECONDARY OUTCOMES:
Change from baseline in other average core gastroparesis symptoms from the Gastroparesis Core Symptom Daily Diary | 12 weeks
  A patient reported daily symptom diary asking patients to rate their nausea on a Likert scale from 0-5 (0=none, 5= very severe). Other symptoms include vomiting, postprandial fullness, early satiety, and abdominal pain
Change from baseline in Patient Assessment of Gastrointestinal Disorders - Symptoms Severity Index (PAGI-SYM) | 12 weeks
  PAGI-SYM is a patient reported outcome that measures specific symptoms of patients with upper gastrointestinal disorders such as gastroparesis, GERD, and dyspepsia on a 0-5 Likert Scale (0=none, 5=very severe).
Change from baseline in Patient Global Impression - Change (PGI-C) | 12 weeks
  A patient reported outcome measuring a patient's rating of overall improvement after treatment on a 7 point scale that includes items "1=very much worse" and "7=very much improved"
Clinician Global Impression - Severity (CGI-S) | 12 weeks
  A clinician reported outcome that measures the clinician's view of the patient's global functioning prior to and after initiating treatment. Symptom severity is measured on a 7 point scale including "1=normal, not at all ill" and "7=among the most extremely ill patients."
Safety and tolerability as measured by spontaneous reporting of adverse events (AEs) | 12 weeks
  Safety will be monitored using clinical measures, vital signs, blood chemistry, hematology, urology, ECGs, and patient reported questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (33):
- United States (33):
  - Vanda Investigational Site, Birmingham, Alabama
  - Vanda Investigational Site, Peoria, Arizona
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Chula Vista, California
  - Vanda Investigational Site, La Jolla, California
  - Vanda Investigational Site, Los Angeles, California
  - Vanda Investigational Site, Maitland, Florida
  - Vanda Investigational Site, Palmetto Bay, Florida
  - Vanda Investigational Site, Tampa, Florida
  - Vanda Investigational Site, Morrow, Georgia
  - Vanda Investigational Site, Wauconda, Illinois
  - Vanda Investigational Site, West Des Moines, Iowa
  - Vanda Investigational Site, Wichita, Kansas
  - Vanda Investigational Site, Louisville, Kentucky
  - Vanda Investigational Site, Marrero, Louisiana
  - Vanda Investigational Site, Chevy Chase, Maryland
  - Vanda Investigational Site, Boston, Massachusetts
  - Vanda Investigational Site, Chesterfield, Missouri
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Brooklyn, New York
  - Vanda Investigational Site, Charlotte, North Carolina
  - Vanda Investigational Site, Raleigh, North Carolina
  - Vanda Investigational Site, Columbus, Ohio
  - Vanda Investigational Site, Huber Heights, Ohio
  - Vanda Investigational Site, Edmond, Oklahoma
  - Vanda Investigational Site, Tulsa, Oklahoma
  - Vanda Investigational Site, Philadelphia, Pennsylvania
  - Vanda Investigational Site, Chattanooga, Tennessee
  - Vanda Investigational Site, Nashville, Tennessee
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Plano, Texas
  - Vanda Investigational Site, San Antonio, Texas
  - Vanda Investigational Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carlin JL, Polymeropoulos C, Camilleri M, Lembo A, Fisher M, Kupersmith C, Madonick D, Moszczynski P, Smieszek S, Xiao C, Birznieks G, Polymeropoulos MH. The Efficacy of Tradipitant in Patients With Diabetic and Idiopathic Gastroparesis in a Phase 3 Randomized Placebo-Controlled Clinical Trial. Clin Gastroenterol Hepatol. 2024 Dec;22(12):2506-2516. doi: 10.1016/j.cgh.2024.01.005. Epub 2024 Jan 17. PMID 38237696
- See also: Study Website — http://www.gpvandastudy.com

DOCUMENTS (2):
  • Study Protocol (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT04028492/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT04028492/SAP_001.pdf